CLINICAL TRIAL: NCT07068269
Title: Effects of Self-management Program of Activity Coping and Education on Quality of Life, Self-efficacy, Exercise Capacity and Anxiety and Depression in Patients With COPD
Brief Title: Self-management Program in Patients With COPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Firasha- REC/RCR&AHS 24/0366
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Chronic Obstr Lung Disease
Keywords: Chronic obstructive pulmonary disease; Self-management program; Activity education and coping
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Self-Management

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Self-Management Program
  Interventions: Other: Self-Management Program
- Group B (Active Comparator): Routine Physical Therapy Exercise
  Interventions: Other: Routine Physical Therapy Exercises

INTERVENTIONS:
Other: Self-Management Program — Week 1: Learn about COPD, practice pursed-lip and diaphragmatic breathing (2-3 sets, 10-15 reps, 2-3x/day), start 5-10 min light walking, conserve energy with frequent rests.
  Week 2: Understand benefits of activity and oxygen use, add seated marches/leg raises, walk 10-15 min, pace activities with rest breaks.
  Week 3: Begin strength exercises (sit-to-stand, wall push-ups, 2 sets of 10), increase walking to 15-20 min, practice relaxation for anxiety.
  Week 4: Focus on nutrition, walk 20-25 min, continue strength work, recognize flare-up signs, create action plan.
  Week 5: Seek social support, walk 25-30 min, add stretching (2-3x/week), track activity daily.
  Week 6: Set SMART goals, maintain daily walking 30 min, review coping strategies, add new activities if desired.
  Arms: Group A
Other: Routine Physical Therapy Exercises — Week 1: Practice pursed-lip and diaphragmatic breathing (2-3 sets, 10-15 breaths, 2-3x/day), start walking 5-10 min (3-5x/week), add gentle upper body stretches (20-30 sec holds, 2-3 reps).
  Week 2: Continue breathing exercises, increase walking slightly each session, maintain stretches 3-5x/week for flexibility.
  Week 3: Keep breathing routines, walk or cycle 15-20 min (4-5x/week), start sit-to-stand strength exercises (2-3 sets of 10-15 reps, 2-3x/week), keep stretching routine.
  Week 4: Maintain breathing drills, increase walking/cycling intensity if tolerated, continue strength work and flexibility exercises.
  Week 5: Keep up breathing exercises, walk/cycle 20-30 min (5x/week), do sit-to-stand exercises (3 sets of 10-15 reps, 3x/week), maintain upper body stretching.
  Week 6: Sustain daily breathing practice, aim for 30 min walking/cycling daily, continue strength and stretch exercises, adjust intensity as needed for long-term progress.
  Arms: Group B

SUMMARY:
The prevalent, preventable, and treatable condition known as chronic obstructive pulmonary disease (COPD) is characterized by ongoing respiratory symptoms and restricted airflow caused by abnormalities of the airways and alveoli. Dyspnea, coughing, sputum production, and exacerbations are among the chronic respiratory symptoms of COPD. The objective of this study is to determine the effects of self-management program of activity coping and education on quality of life, self-efficacy, exercise capacity and anxiety and depression in patients with COPD. People with COPD should be given self-management support, according to national and international recommendations for managing the condition. Hospitalizations, COPD-specific health expenses, and health-related quality of life have all been demonstrated to improve when people with COPD receive interventions that promote self-management.

The study will be randomized clinical trial. Patients age between 45 to 60 years and diagnosed with COPD will be included. The Group A will receive self-management program of activity coping and education for 6 weeks whereas the Group B will receive routine physical therapy for 6 weeks. Pulmonary function testing will be used to evaluate the severity of COPD, St George Respiratory Questionnaire will be used to determine the quality of life, and Self-efficacy of patients will be assessed by COPD Self-efficacy Scale, 6-minute walk test will be used to find the exercise capacity of participants and anxiety and depression will be measured by the Hospital Anxiety and Depression Scale. Data will be analyzed using SPSS version 26.

DETAILED DESCRIPTION:
The prevalent, preventable, and treatable condition known as chronic obstructive pulmonary disease (COPD) is characterized by ongoing respiratory symptoms and restricted airflow caused by abnormalities of the airways (bronchitis) and/or alveoli (emphysema), which are typically brought on by prolonged exposure to harmful particles or gases. Dyspnea, coughing, sputum production, and exacerbations are among the chronic respiratory symptoms of COPD. COPD is a global public health issue and one of the main causes of death and illness, particularly in developing nations. Approximately 30 million Americans are thought to suffer from COPD. Up to half of them are not even aware that they have it. The leading cause of chronic disease, COPD is expected to rank seventh globally in terms of disease burden by 2030. According to estimates, the prevalence of COPD in individuals over 40 is between 4 and 20% worldwide, and 6.3% in Asians. In addition, it is the fourth most frequent reason for hospitalization and the biggest financial burden among chronic illnesses affecting elderly patients.

People with COPD should be given self-management support, according to national and international recommendations for managing the condition. Hospitalizations, COPD-specific health expenses, and health-related quality of life have all been demonstrated to improve when people with COPD receive interventions that promote self-management. Although self-care is implied by the name "self," self-management always entails collaboration with a health care provider, who plays a supportive role. In general, COPD self-management programs are designed to give participants the skills necessary to follow long-term disease-specific medication regimes. The goals of SPACE for COPD, a Self-Management Program of Activity Coping and Education, are to help individuals with COPD manage daily tasks, reduce symptom load, encourage behavior changes that improve health, and improve psychological well-being. Programs for self-management should include physical activity, quitting smoking, managing social interactions, managing medications, and being able to identify and react to symptoms. The SPACE for COPD guidebook, which incorporates both general self-management techniques and disease-specific activities, serves as the framework for the program. Few studies have attempted to assess the cost-effectiveness of self-management programs for individuals with COPD. Some studies simply included the program's expenses. Self-management programs have been shown to be cost-effective in both lowering costs and improving patient outcomes.

This study is significant because it has the potential to concentrate on non-pharmacological interventions, such as self-management programs. A self-management program (SMP) for COPD is a patient-oriented approach that enables the patient to take charge of their condition through appropriate choice making, physical activity, emotional management, education on a continuous basis and encouraging adherence to the treatment plans. Such a program aims at enhancing the quality of life of the patient, and decreasing the frequency of exacerbations while increasing the overall functional ability of the patient. Moreover it reduces hospital admissions and emergency room visits which can alleviate pressure on healthcare systems. Self-management program (SMP) can raise awareness about COPD leading to greater community support. Improved management of symptoms can lead to a more active lifestyle for patients, benefiting overall societal health and productivity.

ELIGIBILITY:
Inclusion Criteria:

* Male and female
* Age 40-65 years
* Participants are eligible for the trial if they have an established diagnosis of COPD as defined by The Global Initiative for Chronic Obstructive Lung Disease (GOLD) criteria

Exclusion Criteria:

* Unable to participate in the exercise component of the SPACE for COPD programme due to neurological, locomotive or psychiatric disability
* Unable to participate in the exercise component of the SPACE for COPD programme due to other comorbidities where exercise would be a contraindication (e.g., unstable angina)

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Pulmonary function testing | Baseline, 3rd Week, 6th Week
St George Respiratory Questionnaire | Baseline, 3rd Week, 6th Week
COPD Self-Efficacy Scale | Baseline, 3rd Week, 6th Week
6-min walk test | Baseline, 3rd Week, 6th Week
Hospital Anxiety and Depression Scale | Baseline, 3rd Week, 6th Week

CONTACTS AND LOCATIONS:
Overall Officials: Danish Hassan, PhD, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehabilitation Clinic, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bourne C, Houchen-Wolloff L, Patel P, Bankart J, Singh S. Self-management programme of activity coping and education-SPACE for COPD(C)-in primary care: a pragmatic randomised trial. BMJ Open Respir Res. 2022 Oct;9(1):e001443. doi: 10.1136/bmjresp-2022-001443. PMID 36253020
- [Background] Gupta N, Agrawal S, Chakrabarti S, Ish P. COPD 2020 Guidelines - what is new and why? Adv Respir Med. 2020;88(1):38-40. doi: 10.5603/ARM.2020.0080. No abstract available. PMID 32153009